CLINICAL TRIAL: NCT06376838
Title: A Randomized, Subject and Evaluator Blinded, Split-face, Pivotal, Multi-injection Clinical Trial to Evaluate the Efficacy and Safety of DLMR01 in Crow's Feet.
Brief Title: To Prove the Non-inferiority of DLMR01 by Evaluating the Injecting Efficacy and Safety DLMR01 and Control for Patients in Crow's Feet
Acronym: dermal filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DEXLEVO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLV-001-02
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Crow's Feet Lines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DLMR01 (Experimental): * one side crow's feet
  * Single dose
  Interventions: Device: DLMR01
- Rejuran (Active Comparator): * one side crow's feet
  * Single Dose
  Interventions: Device: Rejuran

INTERVENTIONS:
Device: DLMR01 — Experimental and Acitve Comparator are applied 1 time to each of crow's feet on both sides of the subject.
  Other Names: Polycaprolactone filler
  Arms: DLMR01
Device: Rejuran — Experimental and Acitve Comparator are applied 1 time to each of crow's feet on both sides of the subject.
  Other Names: Polynucleotide (PN)
  Arms: Rejuran

SUMMARY:
This clinical study is a confirmatory clinical study to prove that the test device, DLMR01, is non-inferior to the control device, Rejuran®, in terms of temporary wrinkle improvement effect on crow's feet and safety. After applying DLMR01, a test device, and Rejuran®, a control device, respectively to wrinkles around the eyes, randomization to compare and evaluate the temporary wrinkle improvement effect and safety of the two clinical study medical devices, subject-evaluator blinding, pair matching, It was designed as a comparative clinical study.

DETAILED DESCRIPTION:
A total of 218 clinical study subjects participated in this clinical study, and the clinical study subjects signed a written informed consent for this clinical study at the screening visit (visit 1), and only if they satisfied various test results and selection/exclusion criteria. Randomly prescribed and applied medical devices for clinical studys (test devices, control devices). A total of 5 visits were scheduled for the subject and visit 1 (screening visit) was conducted within 14 days prior to the first application of the subjects clinical study medical device. Subjects visited the clinical study institution at 2 weeks (visit 3), 4 weeks (visit 4), and 12 weeks (visit 5) after the final application of clinical study medical devices (visit 2) and conducted observation and examination to conduct clinical study. The efficacy and safety of the test medical device were confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. Subjects who voluntarily decided to participate in this clinical trial and provided written consent on the subject's informed consent form were included.
3. Subjects who desired improvement in bilateral crow's feet wrinkles and had a Crow's Feet Grading Scale score of 2 or higher during both rest and maximum smiling were included. It was also required that the crow's feet wrinkles were visually symmetrical on both sides.
4. Subjects who agreed not to undergo any procedures or treatments during the course of the clinical trial that could potentially affect the improvement of periorbital wrinkles, other than the interventions specified in the trial, were included.
5. Subjects who were capable of understanding and following instructions and were available to participate throughout the entire pre-trial period were included.

[Exclusion Criteria]

1. Subjects who had taken anticoagulants (excluding low-dose aspirin, maximum 100mg/day, up to 300mg/day) or non-steroidal anti-inflammatory drugs within 2 weeks from the screening date were excluded.
2. Subjects who had significant liver dysfunction or coagulation abnormalities, or those who needed to take anticoagulants (excluding low-dose aspirin, maximum 100mg/day, up to 300mg/day) during the clinical trial period were excluded.
3. Subjects who had used topical agents (steroids, retinoids - limited to medications, excluding cosmetics) on their face within 1 month prior to the screening date or were planning to use them during the clinical trial period were excluded.
4. Subjects who had undergone invasive laser procedures, deep chemical peels, or any other procedures or surgeries related to wrinkle improvement on their face within 6 months prior to the screening date were excluded.
5. Subjects who had received wrinkle improvement treatments within 6 months prior to the screening date, such as collagen or hyaluronic acid fillers, polyalkylimide fillers, or any other treatments involving the use of injectable substances, were excluded.
6. Subjects who had received wrinkle improvement treatments using calcium hydroxylapatite (CaHA) fillers within 12 months prior to the screening date were excluded.
7. Subjects who had inserted permanent dermal fillers such as softform or silicone for facial augmentation in the facial area were excluded.
8. Subjects who had facial scars that had not been treated for more than 12 months or had scars or marks in the areas where the investigational medical device would be applied were excluded.
9. Subjects who have initiated or applied new wrinkle-preventing medications or cosmetics, including oral or topical formulations with wrinkle prevention effects, within the 3 months prior to their participation in the clinical trial, are excluded.
10. Subjects who currently have skin disorders or wound infections in the facial area were excluded.
11. Subjects with a history of anaphylaxis or severe complex allergies are excluded.
12. Subjects with hypersensitivity or allergic reactions to the components of the product (Polycarprolactone) are excluded.
13. Subjects with a history of hypertrophic scars or keloids are excluded.
14. Subjects who have experienced adverse reactions to EMLA Cream in the past are excluded.
15. Subjects who are drug or alcohol addicts are excluded.
16. Subjects with severe immunodeficiency disorders, including AIDS, or those receiving immunosuppressive therapy are excluded.
17. Subjects with a history of recurrent streptococcal infections are excluded.
18. Subjects with clinically significant disorders affecting the cardiovascular, digestive, respiratory, endocrine, or central nervous systems, or those with significant psychiatric disorders that have had or may have a significant impact on the clinical trial, are excluded.
19. Subjects who have participated in another clinical trial within 1 month prior to the screening date are excluded.
20. Female clinical trial subjects who are of childbearing potential and do not agree to use medically acceptable methods of contraception during the clinical trial period are excluded.
21. Pregnant women, lactating women, and those planning to become pregnant are excluded.
22. Subjects who are deemed by the investigational device to be inappropriate for participation in this clinical trial based on their own judgment are excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Crow's Feet Grading Scale by independent evaluators after 12 weeks of using | independent evaluators after 12 weeks of using the investigational medical device for clinical trials.
  The improvement in wrinkles assessed using the Crow's Feet Grading Scale[The scale grades wrinkles from 0(No wrinkles), 1(Very fine wrinkles),2(Fine wrinkles), 3(Moderate wrinkles), 4(Severe wrinkles)] by independent evaluators after 12 weeks of using the investigational medical device for clinical trials * Wrinkle improvement was evaluated before and after application of clinical study medical devices improved by at least 1 point on the Crow's Feet Grading Scale. It is defined as a case, and the wrinkle improvement rate is the number of wrinkles among the clinical study subjects that can be analyzed, and wrinkles improvement rate is defined as the percentage of wrinkles among analyzable clinical study subjects proportion of selected subjects.

SECONDARY OUTCOMES:
(1) The improvement rate of wrinkles evaluated using the Crow's Feet Grading Scale | 12 weeks of using the investigational medical device for clinical trials, specifically when smiling, was assessed.
  (1) The improvement rate of wrinkles evaluated using the Crow's Feet Grading Scale[The scale grades wrinkles from 0(No wrinkles), 1(Very fine wrinkles),2(Fine wrinkles), 3(Moderate wrinkles), 4(Severe wrinkles)] by independent evaluators after 12 weeks of using the investigational medical device for clinical trials, specifically when smiling, was assessed. * Wrinkle improvement was evaluated before and after application of clinical study medical devices improved by at least 1 point on the Crow's Feet Grading Scale. It is defined as a case, and the wrinkle improvement rate is the number of wrinkles among the clinical study subjects that can be analyzed, and wrinkles improvement rate is defined as the percentage of wrinkles among analyzable clinical study subjects proportion of selected subjects.
(2) The improvement rate of wrinkles assessed using the Crow's Feet Grading Scale by independent evaluators after 2 weeks and 4 weeks of using the medical device both during rest and when smiling was evaluated. | The improvement rate of wrinkles assessed using the Crow's Feet Grading Scale by independent evaluators after 2 weeks and 4 weeks of using the investigational medical device for clinical trials, both during rest and when smiling was evaluated.
  The improvement rate of wrinkles assessed using the Crow's Feet Grading Scale[The scale grades wrinkles from 0(No wrinkles), 1(Very fine wrinkles),2(Fine wrinkles), 3(Moderate wrinkles), 4(Severe wrinkles)] by independent evaluators after 2 weeks and 4 weeks of using the investigational medical device for clinical trials, both during rest and when smiling was evaluated. * Wrinkle improvement was evaluated before and after application of clinical study medical devices improved by at least 1 point on the Crow's Feet Grading Scale. It is defined as a case, and the wrinkle improvement rate is the number of wrinkles among the clinical study subjects that can be analyzed, and wrinkles improvement rate is defined as the percentage of wrinkles among analyzable clinical study subjects proportion of selected subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-ang University Hospital, Seoul, Dongjak-gu, South Korea